CLINICAL TRIAL: NCT03545828
Title: Neurological Prognostication Using Multi-channel Amplitude-integrated Electroencephalographic Monitoring in Cardiac Arrest Patients With Targeted Temperature Management
Brief Title: Multi-channel aEEG in Cardiac Arrest Patients With Targeted Temperature Management
Acronym: MAEGIC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sang Hoon Oh (Other)
Responsible Party: Sponsor-Investigator, Sang Hoon Oh, Associate Professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Other Study IDs: MAEGIC-01
Record Dates: First submitted 2018-04-22; First posted 2018-06-04 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Heart Arrest; Targeted Temperature Management
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Good neurological outcome: CPC 1 and 2 at 6 month after ROSC
  Interventions: Diagnostic Test: Multi-channel aEEG monitoring
- Poor neurological outcome: CPC 3 to 5 at 6 month after ROSC
  Interventions: Diagnostic Test: Multi-channel aEEG monitoring

INTERVENTIONS:
Diagnostic Test: Multi-channel aEEG monitoring — 18 channel aEEG monitoring in comatose TTM-treated patients

SUMMARY:
This study aims to examine the prognostic value of 18 channel amplitude-integrated EEG (aEEG) in comatose cardiac arrest patients The study design is a prospective observational study. Cardiac arrest patients undergoing targeted temperature management (TTM) will participate in the study. Relation of aEEG in each channel with the neurologic outcome at 6 month after return of spontaneous circulation (ROSC) will be evaluated.

DETAILED DESCRIPTION:
Normal trace was defined as continuous cortical activity on the raw EEG scan; in addition, the upper margin of the aEEG scan, referred to as the aEEG maximum, was >10 μ V, and the lower margin of the aEEG scan, referred to as the aEEG minimum, was >5 μ V. The Time from ROSC to normal trace (TTNT, hours) is predictor of neurological outcome in these patients. We will evaluate the prognostic values of TTNTs in all aEEG channels.

ELIGIBILITY:
Inclusion Criteria:

Comatose cardiac arrest TTM treatment Multi channel aEEG monitoring

Exclusion Criteria:

Cerebral origin cardiac arrest Known epilepsy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: TTM treated cardiac arrest patients
Sampling Method: Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to normal trace in each aEEG channel | at day 180
  Normal trace was defined as continuous cortical activity on the raw EEG scan; in addition, the upper margin of the aEEG scan, referred to as the aEEG maximum, was >10 μ V, and the lower margin of the aEEG scan, referred to as the aEEG minimum, was >5 μ V. The Time from ROSC to normal trace (TTNT, hours) is predictor of neurological outcome in these patients. We will evaluate the prognostic values of TTNTs in all aEEG channels.

SECONDARY OUTCOMES:
TTNT threshold for neurologic prognostication in each aEEG channel | at day 180
  Using area under the curve (AUC) of each channel aEEG for neurological outcome, we will determine the best TTNT thresholds for good neurological outcome (CPC 1 to 2) in all aEEG channels.
Alpha delta ratio of each channel aEEG for good neurological outcome (CPC 1 to 2) | at day 180
  The percentage powers in the alpha, theta and delta bands and the ratio of the powers in different frequency bands (i.e., alpha/delta) will be calculated. Finally we will evaluate the prognostic values of these ratios of the different bands.
Comparison of prognostic value between aEEG and various predictors | at day 180
  We will compare the prognostic performances (i.e., sensitivity, specificity, AUC) for poor neurological outcome (CPC 3 to 5) between EEG and these predictors.

CONTACTS AND LOCATIONS:
Overall Officials: Sang Hoon Oh, Study Director — Seoul St. Mary's Hospital
Locations (1):
- Seoul St. Mary's hospital, Seoul, South Korea